CLINICAL TRIAL: NCT03615963
Title: Aortic Root Distensibility And Stiffness Assessed By Echocardiography As Predictors Of Coronary Artery Lesion Severity In Coronary Artery Patients Undergoing Coronary Angiography
Brief Title: Aortic Stiffness and Distensibility as Predictor to Severity of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HSAnwar, Principal investigator, Assiut University
Other Study IDs: Aortic stiffness
Record Dates: First submitted 2018-07-05; First posted 2018-08-06 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Echocardiography; Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal: patient complains of anginal chest pain but coronary angiography is normal
  Interventions: Diagnostic Test: echocardiography and coronary angiography
- coronary artery disease: patient complains of chest pain with coronary angiography showing atherosclerotic plaques causing luminal obstruction
  Interventions: Diagnostic Test: echocardiography and coronary angiography

INTERVENTIONS:
Diagnostic Test: echocardiography and coronary angiography — transthoracic echocardiography will be done for all subjects to measure aortic stiffness and elaticity then coronary angiography was used to differentiate between normal subjects and who have coronary artery disease

SUMMARY:
Assess the relationship of Aortic root distensibility and stiffness with the extent of coronary artery disease as assessed by SYNTAX score compared to a matched cohort of patients with normal coronary angiography

DETAILED DESCRIPTION:
Cardiovascular disease leading cause of death, resulting in a number of annually deceased people higher than from any other. The great incidence of cardiovascular diseases in the world spurred the search for new solutions to enable an early detection of pathological processes The early detection based in multi-parameters of pathological condition is the key to the patient survival .The arterial stiffness is the first vessels modification, responsible for several pathological processes, which can lead to cardiovascular diseases.

The normal aging process is associated with an increase in vascular stiffness which is accelerated by atherosclerosis, hypertension, and diabetes mellitus. Several studies have revealed that increased aortic stiffness is a risk factor for cardiovascular diseases and also is a predictor of cardiovascular morbidity and mortality.

Interest in arterial stiffness waned in the early 1900s with the advent of the sphygmomanometer, which offered a quantitative measure of blood pressure and risk prediction .

Another factor is Aortic distensibility which is a measurement of vascular elasticity, and reflects the stiffness of the aorta . Aortic distensibility is markedly decreased in patients with known coronary artery disease . and is inversely proportional to the severity of Coronary artery disease .

Two-dimensional and tissue Doppler imaging derived parameters of ascending aorta have been found to be abnormal, indicating increased Aortic stiffness and impaired Aortic distensibility in subjects with coronary artery disease, hypertension, and diabetes mellitus. However, the direct correlation of Aortic stiffness with Coronary artery disease is hard to examine as most of these patients are old and have comorbidities such as hypertension, So Investigation of these parameters should be done in patients who are normotensive as most of these patients do not have confounding factors that increase Aortic stiffness.

Although the relationship between Aortic distensibility and Aortic stiffness and atherosclerosis is well known , the possible relation between them and the extent and complexity of coronary artery disease. as assessed using SYNTAX score has not been clearly determined yet.

The SYNTAX score is a lesion-based angiographic scoring system originally devised to grade the complexity of coronary artery disease.

. It is related to adverse cardiovascular events and predicts mortality and morbidity in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* all patients suspected to have coronary artery disease

Exclusion Criteria:

* -Hypertension( SBP>140mmhg or DBP>90mmhg)
* Previous coronary stenting
* Previous CABG
* Renal diseases.
* Decompensated liver disease.
* Connective tissue diseases.
* Aortic valve disease ( more than mild aortic stenosis or regurgitation)

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient suspected to have coronary artery disease based on clinical date will underwent echocardiography to measure aortic root stiffness and elasticity then coronary angiography will be done to differentiate normal and coronary artery disease .
  then aortic root stiffness and elasticity will be compared between the two groups.
  is aortic root stiffness and elasticity can predict coronary artery disease and its severity
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
compare aortic stiffness and elasticity in normal subjects and patient with coronary artery disease | 1 hour
  aortic stiffness by echocardiography ⊿P=Ps-Pd mmHg. ⊿D=As-Ad cm. local arterial stiffness can be calculated using the following formula: Aortic distensibility (AD) cm2/dyn= (2x⊿D)/((Adx⊿p)) Aortic stiffness index(SI)= ln (Ps/Pd)/(⊿D/Ad) no units ln is the natural logarithm Arterial strain = (⊿D)/Ad no units The elastic modulus E(p) = (⊿P)/Strain ( mmHg/cm) tissue doppler imaging (TDI) The TDI of expansion peak velocity during systole (SAo) and early (EAo) and late (AAo) diastolic peak velocities (m/s)are obtained
  then coronary angiography will be done to differentiate the 2 groups into normal and others have coronary artery disease using Syntax score( SS) Patients were divided into three tertiles: SS LOW ≤22 22< SSMID ≤32 SS HIGH >32

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Demitry, Study Director — Assiut University
Locations (1):
- Helen Sami Anwar, Asyut, Egypt

REFERENCES:
- [Background] Wilkinson IB, Cockcroft JR, McEniery CM. Aortic stiffness as a cardiovascular risk predictor. BMJ. 2015 Jul 14;351:h3764. doi: 10.1136/bmj.h3764. No abstract available. PMID 26173600
- [Background] Wang F, Ye P, Luo L, Xiao W, Qi L, Bian S, Wu H, Sheng L, Xiao T, Xu R. Association of serum lipids with arterial stiffness in a population-based study in Beijing. Eur J Clin Invest. 2011 Sep;41(9):929-36. doi: 10.1111/j.1365-2362.2011.02481.x. Epub 2011 Feb 14. PMID 21314825
- [Background] Zhang YJ, Iqbal J, Campos CM, Klaveren DV, Bourantas CV, Dawkins KD, Banning AP, Escaned J, de Vries T, Morel MA, Farooq V, Onuma Y, Garcia-Garcia HM, Stone GW, Steyerberg EW, Mohr FW, Serruys PW. Prognostic value of site SYNTAX score and rationale for combining anatomic and clinical factors in decision making: insights from the SYNTAX trial. J Am Coll Cardiol. 2014 Aug 5;64(5):423-32. doi: 10.1016/j.jacc.2014.05.022. PMID 25082573